CLINICAL TRIAL: NCT01986231
Title: The Effect of Repeated Doses of Subcutaneous Glucagon on Hepatic Glycogen Stores in Persons With Type 1 Diabetes
Brief Title: Safety Study of Repeated Doses of Glucagon on Animal Starch in the Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, W. Kenneth Ward, Senior Scientist, Legacy Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00006947
Record Dates: First submitted 2013-11-05; First posted 2013-11-18 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; insulin; glucagon; glycogen; MRS
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label Glucagon (Experimental): Subjects will receive 8 doses of glucagon, each dose will be 2.0 mcg per kg.
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — Subjects will receive 8 doses of glucagon, each dose will be 2.0 mcg per kg. Glucagon will be reconstituted immediately prior to administration and each dose will be administered subcutaneously via syringe/needle. The first glucagon dose is at hour 17, second at hour 22, third at hour 24, fourth at hour 27, fifth at hour 29, sixth at hour 31, seventh at hour 33, eighth at hour 35.
  Other Names: GlucaGen

SUMMARY:
The purpose of this study is to learn if giving multiple doses of a hormone called glucagon can cause a major decrease in liver glycogen (animal starch). Glucagon is currently approved by the Food and Drug Administration to be given as a large dose to treat severe low blood sugar. Our group is studying whether glucagon can be given in repeated small doses to prevent hypoglycemia.

DETAILED DESCRIPTION:
Hypoglycemia remains a barrier to optimal glucose control, which is necessary to prevent diabetes-related complications including eye, kidney, and nerve diseases. Despite treatment advances such as insulin pump therapy and continuous glucose monitoring, hypoglycemia remains a concern, even when insulin is given in a closed-loop system. A closed-loop system consists of a glucose-measuring device, from which data are collected and entered into an algorithm, which in turn controls insulin delivery. The difficulty of delivering regular or analog insulin in such a manner is related to its slow onset and prolonged effect when delivered subcutaneously. Until a more rapidly-acting insulin preparation is available, discontinuation of subcutaneous insulin during impending hypoglycemia, with any algorithm, may be insufficient to prevent hypoglycemia.

Glucagon, a hormone secreted from the alpha cells of the normal endocrine pancreas, rapidly raises circulating glucose levels within minutes via glycogenolysis, even when given subcu-taneously. Glucagon is approved for use as a parenteral injection for treatment of severe hypoglycemia. Our group has successfully completed studies in humans using a closed-loop system that delivers insulin (in a nearly continuous fashion) to prevent and treat hyperglycemia as well as glucagon (intermittently) to prevent and treat hypoglycemia.

However, it is unknown whether or not repeated doses lead to hepatic glycogen depletion, which would increase the risk of a severe hypoglycemic episode. 13C MRS (magnetic resonance spectroscopy) has been successfully used to quantify hepatic glycogen in a non-invasive fashion. We are proposing to use 13C MRS to compare glycogen stores in subjects with type 1 diabetes after a period without glucagon vs after a period of repeated glucagon dosing. The comparisons will be made when glycogen stores should be replete (after a lunch meal) and when glycogen stores should be lower (after an overnight fast). If repeated doses of glucagon do cause glycogen depletion, then we would revise our dosing strategy in the closed-loop system and/or consider alternative methods for preventing hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed for at least 6 months
* Current usage of subcutaneous insulin pump treatment
* Age 18-65 years
* HbA1c of 5.5 - 7.7% at screening visit
* BMI 18-35 kg/m2
* Willingness to follow all study procedures, including attending all clinic visits
* Willingness to sign informed consent and HIPAA documents

Exclusion Criteria:

* Pregnancy or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test.
* Renal insufficiency (serum creatinine of 2.0 mg/dL or greater).
* Serum ALT or AST equal to or greater than 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as a serum albumin of less than 3.3 g/dL; or serum bilirubin of over 2.
* Hematocrit of less than or equal to 34%.
* Congestive heart failure, NYHA class II, III or IV.
* Coronary artery or cerebrovascular disease.
* Active foot ulceration.
* Active alcohol abuse, substance abuse, or severe mental illness (as judged by the principal investigator).
* Active malignancy, except basal cell or squamous cell skin cancers.
* Major surgical operation within 30 days prior to screening.
* Seizure disorder (epilepsy).
* Contraindication to an MRI scan, including having metallic splinters in the eye, a cardiac pacemaker, defibrillator, or any other ferromagnetic or electronically charged implanted device, or ferromagnetic clip(s) in the central nervous system.
* Currently administration of oral or parenteral corticosteroids.
* Use of an investigational drug within 30 days prior to screening.
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* History weight loss of ≥ 5 lbs over the prior month.
* Weight ≥ 300 lbs.
* Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
* Any reason the principal investigator deems exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W Kenneth Ward, MD, Principal Investigator — Legacy Health System
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Castle JR, El Youssef J, Bakhtiani PA, Cai Y, Stobbe JM, Branigan D, Ramsey K, Jacobs P, Reddy R, Woods M, Ward WK. Effect of Repeated Glucagon Doses on Hepatic Glycogen in Type 1 Diabetes: Implications for a Bihormonal Closed-Loop System. Diabetes Care. 2015 Nov;38(11):2115-9. doi: 10.2337/dc15-0754. Epub 2015 Sep 4. PMID 26341131

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Glucagon: Subjects will receive 8 doses of glucagon, each dose will be 2.0 mcg per kg. Glucagon will be reconstituted immediately prior to administration and each dose will be administered subcutaneously via syringe/needle. The first glucagon dose is at hour 17, second at hour 22, third at hour 24, fourth at hour 27, fifth at hour 29, sixth at hour 31, seventh at hour 33, eighth at hour 35.
  Glucagon: Subjects will receive 8 doses of glucagon, each dose will be 2.0 mcg per kg. Glucagon will be reconstituted immediately prior to administration and each dose will be administered subcutaneously via syringe/needle. The first glucagon dose is at hour 17, second at hour 22, third at hour 24, fourth at hour 27, fifth at hour 29, sixth at hour 31, seventh at hour 33, eighth at hour 35.
Period: Overall Study
Arm/Group | Open-Label Glucagon
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Glucagon
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Assess Difference in Hepatic Glycogen Measured in the Fasting State Before vs. After Repeated Glucagon Administration
Description: The mean difference in estimated hepatic glycogen will be assessed using Carbon 13 Magnetic Resonance Spectroscopy before vs. after glucagon administration in the fasting state.
Time Frame: Baseline and 41 hours
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Open-Label Glucagon
Number analyzed (Participants) | 11
g/L | 6.5 (4.5)

2. Secondary Outcome: Assess Difference in Hepatic Glycogen Measured in the Fed State Before vs. After Repeated Glucagon Administration
Description: The mean difference in estimated hepatic glycogen will be assessed using Carbon 13 Magnetic Resonance Spectroscopy before vs. after glucagon administration in the fed state.
Time Frame: Baseline and 41 hours
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Open-Label Glucagon
Number analyzed (Participants) | 11
g/L | 10.6 (7.7)

ADVERSE EVENTS:
Arm/Group | Open-Label Glucagon
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Glucagon (N=12)
headache (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
lightheadedness (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes